CLINICAL TRIAL: NCT06945068
Title: An Open-label Study Evaluating the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, Immunogenicity, and Preliminary Clinical Activity of GB261 in Patients With Refractory Seropositive Systemic Lupus Erythematosus
Brief Title: An Open-label Study of GB261 in Refractory Seropositive Systemic Lupus Erythematosus
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Qiubai Li, Director, Head of Department of Rheumatology and Immunology, Principal Investigator, Professor, Wuhan Union Hospital, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UHCT250170
Record Dates: First submitted 2025-04-10; First posted 2025-04-25 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Systemic Lupus Erythematosus (SLE)
Keywords: Systemic Lupus Erythematosus; GB261
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GB261 intravenous intervention (Experimental): GB261 will be administered by intravenous infusion, including 3 escalating dose levels and subsequent dose expansion. Timepoint of treatment: Day 1, Day 8 and Day 15. Anticipated enrollment: 9-18 participants in Dose Escalation group; 10 participants in Dose Expansion group.
  Interventions: Biological: GB261

INTERVENTIONS:
Biological: GB261 — GB261 will be dosed according to the assigned group.

SUMMARY:
The purpose of the study is to evaluate the safety and efficacy of CD20xCD3 T-cell engager (GB261) in patients with refractory seropositive systemic lupus erythematosus.

DETAILED DESCRIPTION:
B cells play an important role in the pathogenesis of systemic lupus erythematosus (SLE). CD20 is a transmembrane receptor that is highly expressed on approximately 95% of B lineage cells. The use of anti-CD20 for B cell depletion represents a significant breakthrough in the treatment of B-cell-mediated autoimmune diseases. GB261 is a novel CD20/CD3 bispecific TCE that is designed to have very low affinity for CD3 and high affinity for CD20 to enable efficient T cell-mediated killing while minimizing risk of cytokine release syndrome (CRS). GB261 has shown promising safety and anti-tumor activity in a Phase 1/2 study in patients with relapsed/refractory B-cell non-Hodgkin lymphoma and chronic lymphocytic leukemia. GB261 offers a promising mechanism of action for SLE. This study aims to assess the safety, tolerability, PK, pharmacodynamics (PD), immunogenicity, and preliminary clinical activity of GB261 administered in patients with SLE. Patients will be invited to participate in the study, to receive GB261 intravenous infusion and monitored from the first dose of GB261 until Week 52.

ELIGIBILITY:
Inclusion Criteria:

1. 18 to 75 years old at the time of signing the informed consent form (ICF)
2. Diagnosis of SLE according to the 2019 American College of Rheumatology (ACR), European Alliance of Associations for Rheumatology (EULAR) classification criteria
3. 3. Positive for 2 out of 3 antibodies at Screening: a. Anti-dsDNA; b. Anti-Smith antibodies; c. Antinuclear antibody (ANA) titer ≥1:80
4. Active SLE disease
5. Inadequate response
6. Current and stable use of some medication up to Day 1
7. Current and stable use of some medication must be discontinued ≥1 week prior to Day 1

Additional Inclusion Criteria for SLE with Active LN

SLE patients with active LN are eligible to be included in the study only if all of the following additional criteria apply:

1. Active, biopsy-proven, proliferative LN Class III or IV according to the 2018 International Society of Nephrology/Renal Pathology Society criteria
2. Inadequate response
3. Stable angiotensin-converting enzyme inhibitors/angiotensin receptor blockers for at least 4 weeks prior to Screening

Exclusion Criteria:

1. Inadequate clinical laboratory parameters at Screening:
2. Patients will be excluded if they are known to have active infection
3. Receipt of or inability to discontinue any excluded therapies
4. Receipt of live vaccine within 4 weeks prior to Screening
5. Presence of any concomitant autoimmune disease
6. Active or known history of catastrophic anti-phospholipid syndrome (APS)
7. APS or thrombotic event not adequately controlled by anticoagulation therapy
8. History of progressive multifocal leukoencephalopathy
9. History of primary immunodeficiency or a hereditary deficiency of the complement system
10. Central nervous system (CNS) disease
11. Presence of 1 or more significant concurrent medical conditions per investigator judgment
12. Have a diagnosis or history of malignant disease within 5 years prior to Screening
13. Serious mental illness, alcohol or drug abuse, dementia, or any other condition that would impair the patient's ability to receive the planned treatment or to understand informed consent at the study site as determined by local practice
14. Inability to comply with protocol-mandated requirements
15. History of severe allergic or anaphylactic reactions to mAb therapy (or recombinant antibody-related fusion proteins) or any constituents of study drug.
16. History of or planned organ transplant and/or autologous or allogeneic hematopoietic stem cell transplantation for the duration of the study.
17. Major surgery requiring use of general anesthesia within 12 weeks prior to Screening or planned or expected major surgery during the study period (from Screening to patient's last visit).
18. Any serious medical condition or abnormality on clinical laboratory testing
19. Women who are pregnant or breastfeeding.
20. Sexually active male patients who do not agree to refrain from donating semen

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability | Baseline to Month 12
  Incidence and severity of TEAEs through end of study. Cytokine release syndrome (CRS) and immune effector cell-associated neurotoxicity syndrome (ICANS) are graded by ASTCT criteria, other AEs are assessed by CTCAE V5.0 criteria

SECONDARY OUTCOMES:
Pharmacokinetics of GB261 | Baseline to Month 12 (Day1-4, 8-11, 15-18, 22, 29, 36 Week 8, 52)
  PK profiles and parameters, including Peak Plasma Concentration (Cmax), derived for GB261
Pharmacokinetics of GB261 | Baseline to Month 12 (Day1-4, 8-11, 15-18, 22, 29, 36 Week 8, 52)
  PK profiles and parameters, including Area under the plasma concentration versus time curve (AUC), derived for GB261
Pharmacokinetics of GB261 | Baseline to Month 12 (Day1-4, 8-11, 15-18, 22, 29, 36 Week 8, 52)
  PK profiles and parameters, including Time to Maximum Concentration (Tmax) derived for GB261
Pharmacokinetics of GB261 | Baseline to Month 12 (Day1-4, 8-11, 15-18, 22, 29, 36 Week 8, 52)
  PK profiles and parameters, including Half-life (t½), derived for GB261

OTHER OUTCOMES:
Pharmacodynamics of GB261 | Baseline to Month 12(Screening, Day1, Day 8, 15, 22, 29, 36, Week 8, 16, 24, 36, 52)
  Changes from baseline in CD19+ B cells counts.
Pharmacodynamics of GB261 | Baseline to Month 12(Screening, Day1, Day 8, 15, 22, 29, 36, Week 52)
  Changes from baseline in inflammatory cytokines.
Immunogenicity of GB261 | Baseline to Month 12 (Day1, Day 8, 15, 22, 29, 36, Week 8, 12, 16, 24, 52)
  Proportion of patients with ADAs before and after treatment
Patient-reported outcomes | Baseline to Month 12 (Screening, Day1, Day 8, 15, 29, Week 8, 12, 16, 24, 36, 52)
  Change from baseline through Week 52 in Health Assessment Questionnaire - Disability Index (HAQ-DI). Range [0, 3], higher score represents more severe disability.
Effect on affected tissues | From the baseline to Month 12 (Screening and Day 29).
  Changes from baseline in cellular composition. Lymph node biopsy or Bone marrow biopsy.
Clinical activity of GB261 | Baseline to Month 12 (Screening, Day1, Day 8, 15, 29, Week 8, 12, 16, 24, 36, 52)
  Change from baseline in Systemic Lupus Erythematosus Disease Activity Index 2000 (SLEDAI-2K). Range[0, 105], higher score represents worse disease activity

CONTACTS AND LOCATIONS:
Overall Officials: Qiubai Li, Professor, Principal Investigator — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Locations (1):
- Wuhan Union Hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No